CLINICAL TRIAL: NCT04472013
Title: Systematic Assessment of SARS-CoV-2 Neurotropic Capacity in Modestly and Critically Ill Patients, and Patients Who Died From COVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Botnar Research Centre for Child Health (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-01503; ch20Hutter
Record Dates: First submitted 2020-07-14; First posted 2020-07-15 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2022-11

CONDITIONS: COVID-19 Disease
Keywords: SARS-CoV-2; neurotropism of SARS-CoV-2; microglia; CODEX (high dimensional microscopy) analysis
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biological material is appropriately stored in a restricted area only accessible to authorized personnel. The acquired fluids of lumbar puncture, blood withdrawal and autopsy (in case of death) are going to be frozen at -80° C and stored at Department of Biomedicine, University Hospital of Basel. Biological material in this project is not identified by participant name but by a unique participant number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection from lumbar puncture — Cerebro spinal fluid (CSF) will be acquired by lumbar puncture and sent for routine analysis including CSF chemistry, cytology and microbiology. Targeted CSF proteomics using OLINK Proximity Extension Assay (PEA) technology to assess a potential CNS-contribution of the disease will be performed.
Other: Data collection from blood draw — Plasma samples will be acquired for plasma cytokine proteomics using CyTOF (mass cytometry analysis) technology.
Other: CNS magnetic resonance imaging (MRI) imaging — 3Tesla magnetic resonance imaging (MRI) will be performed to document early/manifest encephalitic changes in COVID-19 patients.
Other: Microscopy of defined brain regions on autopsy specimens — High dimensional, microglia-centric CODEX fluorescent microscopy of defined brain regions on autopsy specimens will be acquired from medulla oblongata, cortex, cerebellum, and olfactory bulb. A brain-specific CODEX panel for the assessment of the immune microenvironment was implemented, with inclusion of a wide array of myeloid/microglia markers, T-cell markers, and a few neuronal markers. All the antibodies have been validated and tested in formalin-fixed tissues of different zones of glioblastoma tumors including invading tumor periphery. The Panel will be modified to include the viral entry receptors, CD147, ACE2 and TMPRSS2. Presence of SARS-CoV-2 virus particles will be assessed by qPCR, andMultiplexed Ion Beam Imaging (MIBI) technology will be used to visualize tropism of virus to specific cellular brain compartments.

SUMMARY:
This study is to analyze the microglia reaction or direct neurotropic effects of CNS COVID-19 in pathogenesis and brain stem dysfunction in critically ill patients. A microglia-focused, brain-specific 50+ marker CODEX panel is used to assess the neuroinflammatory microenvironment in specific brain regions of deceased COVID-19 patients. The peripheral (cerebrospinal fluid and peripheral blood) cytokine response to SARS-CoV-2 is investigated in regard to CNS affection and consecutive blood brain barrier disruption leading to braininherent neuroinflammatory reactions

DETAILED DESCRIPTION:
This study is to analyze the microglia reaction or direct neurotropic effects of CNS COVID-19 in pathogenesis and brain stem dysfunction in critically ill patients. A microglia-focused, brain-specific 50+ marker CODEX panel is used to assess the neuroinflammatory microenvironment in specific brain regions of deceased COVID-19 patients. The peripheral (cerebrospinal fluid and peripheral blood) cytokine response to SARS-CoV-2 is investigated in regard to CNS affection and consecutive blood brain barrier disruption leading to braininherent neuroinflammatory reactions. Primary endpoints of this project are the multidimensional integration of the analysis from the procedures described above and assessment of the correlation between the gained clinical data (MRI, mental/neurological state), the body fluid proteomic and mass-cytometric analysis (CSF and Plasma proteomics, peripheral blood mass cytometry) and the CODEX analysis of defined brain regions on autopsy specimens.

Non-critically ill COVID-19 patients and critically ill COVID-19 patients needing mechanical ventilation at the ICU are included. Autopsy specimens from medulla oblongata, cortex, cerebellum and olfactory bulb are investigated, including only tissue samples, which have been submitted to the Institute of Pathology, University Hospital Basel.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive tested

Exclusion Criteria:

* COVID-19 negative tested
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 non-critically ill COVID-19 patients from the inpatient ward, and 20 critically ill COVID-19 patients needing mechanical ventilation at the ICU. Recruitment takes places at University Hospital of Basel and the Kantonsspital Baselland Liestal.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
MRI imaging data | Project duration for each patient takes 1 hour for the MRI at baseline
  Comparison of lesions from patients that are neurologically affected to non-affected individuals in terms of CNS involvement to describe encephalitic changes due to COVID-19 infection.
Proteomic analysis | 10 minutes for blood draw at baseline
  Description of proteomic biomarkers (CSF and Plasma) in comparison with control reference sample.
Peripheral blood leukocyte Cytof Mass Cytometry Analysis for cell population frequency | 10 minutes for blood draw at baseline
  Mass cytometry will be performed form peripheral blood mononuclear cells to count cell population frequency.
CODEX (high dimensional microscopy) workflow analysis of defined regions on brain autopsy specimens | at baseline
  In situ distribution assessment of marker expression (CD147 protein, ACE2 protein, Transmembrane protease serine subtype 2 (TMPRSS2))

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Hutter, Prof. Dr. med., Principal Investigator — Neurosurgery, University Hospital Basel
Locations (1):
- Neurosurgery, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Result] Etter MM, Martins TA, Kulsvehagen L, Possnecker E, Duchemin W, Hogan S, Sanabria-Diaz G, Muller J, Chiappini A, Rychen J, Eberhard N, Guzman R, Mariani L, Melie-Garcia L, Keller E, Jelcic I, Pargger H, Siegemund M, Kuhle J, Oechtering J, Eich C, Tzankov A, Matter MS, Uzun S, Yaldizli O, Lieb JM, Psychogios MN, Leuzinger K, Hirsch HH, Granziera C, Probstel AK, Hutter G. Severe Neuro-COVID is associated with peripheral immune signatures, autoimmunity and neurodegeneration: a prospective cross-sectional study. Nat Commun. 2022 Nov 9;13(1):6777. doi: 10.1038/s41467-022-34068-0. PMID 36351919
- See also: Severe Neuro-COVID is associated with peripheral immune signatures, autoimmunity and neurodegeneration: a prospective cross-sectional study — http://doi.org/10.1038/s41467-022-34068-0